CLINICAL TRIAL: NCT05094219
Title: Disease Burden of Parkinson's Disease in Hong Kong
Brief Title: Disease Burden and Cost Consequence of Falls Among Individuals With Parkinson's Disease in Hong Kong: A Prospective Cost-utility Analysis
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other); The University of Hong Kong (Other); Parkinson's Disease Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: HMRF_K-ZC5K
Record Dates: First submitted 2021-10-17; First posted 2021-10-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
Keywords: Falls; Cost; Disease burden; Economic evaluation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group: Patients with a confirmed diagnosis of Parkinson's disease will be followed up for 12 months from the date of enrollment.
  Interventions: Other: No intervention will be offered

INTERVENTIONS:
Other: No intervention will be offered — No intervention will be offered

SUMMARY:
Objective: Estimate the cost of disease and falls among people with Parkinson's disease living in Hong Kong.

Design: Prospective cost-utility analysis (base year 2021) with one baseline and two follow-up assessments at 6 months and 12 months Participants: Community-dwelling participants with Parkinson's disease of both genders of any age.

Intervention: Nil Outcome measures: Self-reported questionnaires will be used to obtain information about the healthcare utility. In addition, the number of falls, the severity of Parkinson' disease assessed using the MDS-Unified Parkinson's Disease Rating Scale, level of disability using the Hoehn and Yahr scale, balance using the Mini Balance Evaluation Systems Test and Activities-specific Balance Confidence (ABC) scale, risk of falls using Falls Efficacy Scale International and quality of life using the Short-form Health survey (SF-36) will be assessed. Predictors of cost include fall frequency, balance status, disease severity, level of disability, quality of life, and duration of disease.

Analysis: A multiple regression analysis will be conducted to determine which predictor (independent variable) influence the overall cost. The level of statistical significance (α) will be set at p<0.05. A Tornado plot will be constructed for the individual items of both direct and indirect cost having the minimum and maximum range set at the 25th and 75th percentile. Two-way analysis of variance (ANOVA) will assess the differences in healthcare cost among frequent, in-frequent and non-fallers. Spearman's or Pearson correlation coefficient will assess correlations between quality of life and healthcare cost; disease severity and healthcare cost; falls frequency and healthcare cost.

Benefits to healthcare and health Cost-estimation highlights information required to enhance the health care service for the target population. Through a similar study among patients with cerebellar ataxia, our team demonstrated specific challenges that need additional support from the policy-makers such as employment following disability, visits to specialists, home-care, and community participation for people with cerebellar ataxia in Hong Kong. This study will highlight the strength and weakness of the current healthcare system to people of Hong Kong with Parkinson's disease, this will inform the challenges for the healthcare requiring additional attention which in turn will have a beneficial impact on the future service.

DETAILED DESCRIPTION:
Introduction Parkinson's disease is a complex neurodegenerative disorder resulting in a range of complications for both the individual and their families eventually leading to increased burden to the healthcare system.1 Reports from the year 2012 indicated 13,000 (0.186%) people in Hong Kong living with Parkinson's disease 2 and a recent global estimate in 2016 indicates 6.1 million people.3 Postural instability, freezing of gait and poor balance resulting in frequent falls are hallmarks of Parkinson's disease 4. Falls constitute the greatest health and injury risk related to people living with Parkinson's disease. 5, 6

The burden of falls:

Forty-six per cent of people with Parkinson's disease fall at least once every 3 months.7 A recent report suggests 35% to 90% of people with Parkinson's disease fall at least once after being diagnosed with the disease, with an average falls rate of 61%, with about 39% of these being recurrent.8 The sequelae of accidental falls are associated with a decrease in quality of life, increase in caregiver's burden, hip fractures, an increase in motor impairment, decreases in mobility and an increase in disease severity. It is therefore imperative to prevent falls in people with PD.

Falls prevention framework in Hong Kong:

The Elderly Health Service of the Department of Health, HKSAR has published the framework for falls prevention and management.12 The current framework for preventive care for older adults in Hong Kong emphasises fall prevention through physical exercise and pain management. Physical exercises for falls management often include balance training as well as improving muscle strength and mobility. However, these frameworks are for older adults in general. These recommendations have not been developed for individuals with Parkinson's disease, specifically, who both (a) are arguably at more risk of falls and related injuries, and (b) likely require special adaptations for common treatments, given their high rates of disability. Thus, there is a critical need for a similar framework for people with Parkinson's disease in Hong Kong. The proposed study is a necessary first step in the development of such a framework and would provide data that would inform such a framework for people with Parkinson's disease.

Aims and hypothesis

The overall aim of this proposal is to estimate the economic burden of Parkinson's disease from a societal perspective of Hong Kong. To address this aim the following specific objectives are set:

Objective 1: Estimate the total cost and determine the degree to which each direct and indirect cost items influence the total cost per 12 months in Hong Kong.

Objective 2: Assess the impact of falls frequency, balance status, disease severity, level of disability, quality of life, and duration of disease on the overall healthcare cost among people with Parkinson's disease.

Objective 3: Estimate the frequency of falls and compare the cost consequence due to falls between frequent, in-frequent and non-fallers with Parkinson's disease in Hong Kong for 12 months.

Objective 4: Establish the correlation between disease severity, falls frequency and cost.

Methodology Subjects: community-dwelling participants with a confirmed diagnosis of Parkinson's disease of both genders of any age and who are residing in Hong Kong. The data will be collected via the Hong Kong Parkinson's Disease Foundation (attached support letter). In addition, advertisement flyers for recruitment will be posted at the Neighbourhood Advice-Action Council (NAAC) and Caritas (attached support letter) spread across the three districts of HK (i.e., Hong Kong Island, Kowloon and the New Territories). Those who give written consent to participate and are willing to involve and complete a cost questionnaire over 12 months period from the day for enrollment will be included. Volunteers will be excluded if they (1) are wheelchair-bound or bed-ridden, (2) have atypical Parkinson's syndrome and (3) other associated major illness such as stroke. All participants will be assessed during the 'on' phase of the levodopa treatment cycle.

Methods This methodology is in line with the standard guidelines for cost estimation. The ethics approval will be obtained from the Human Subjects Ethics Committee of the Hong Kong Polytechnic University. This trial will be registered with the Clinical Trials Registry or the Open Science. Self-reported questionnaires will be to obtain information about the healthcare utility and the cost will be estimated for the base year 2021 in Hong Kong Dollars (HKD). A baseline assessment will record the demographic data, while the disease severity, fear of falls and quality of life will be assessed using standardized questionnaires and outcome measures. The participants will be instructed to complete the cost questionnaire every week over the 12 months follow up period.

Study design This is a prospective cost-utility analysis with one baseline and two follow-up assessments at 6 months and 12 months.

Sample size: 90 participants with Parkinson's disease. Demographic data: include age, age during disease onset, caregiver information, education level, past medical history, ambulatory status, employment status, housing status and falls history.

Cost data: The participant's healthcare utility will be recorded using an online-based self-reported questionnaire. Printed versions of the questionnaires will be handed to participants with limited access to the internet. The cost-of-illness (COI) analysis also known as the burden of disease (BOD) will be done for this estimation. The COI analysis takes into consideration the impact of the health outcomes on the country, specific regions, communities, and as well as individuals. COI evaluates the morbidity in relation to the decrease in health status and quality of life (QoL), as well as the financial aspects including direct and indirect expenditures that result from premature death, disability or injury.

Cost estimation:

Both direct and indirect cost using the self-reported questionnaires will be recorded in both English and Chinese languages. The following criteria were used to choose the individual items under direct and indirect costs: relevance to Parkinson's disease, relevance to falls and consequences of falls, how quantifiable the items are, based on the commonly estimated items in similar economic, and to the extent to which the item reflects and impacts the quality of life of people with Parkinson's disease.The direct cost items and some of the indirect cost items will be obtained in physical units and not the actual money spent. The physical units will then be converted into monetary units using the human capital method.

Direct cost: Direct costs refers to those expenditures that are directly related to the intervention for the health condition. In this study, the cost items include: (a) inpatient care (general hospital admission due to Parkinson's disease, or falls or other associated problems, visit emergency care for Parkinson's disease or falls of other associated problems, admission at the Intensive care unit), (b) out-patient care (visit to the general practitioner for Parkinson's disease or falls or other associated problems, visit Traditional Chinese Medicine for Parkinson's disease or falls or other associated problems), (c) drugs, (d) rehabilitation, (e) walking aids, and (f) miscellaneous including surgery. The charges for these cost items are derived from the unsubsidized rate for healthcare in Hong Kong published by the Hospital Authorities.

Indirect cost: Indirect cost refers to the expense that is related to the consequence of the disease such as work absenteeism, early retirement, reduced work productivity. In this study, indirect costs include: (a) costs for hiring caregivers, (b) home modification, (c) productivity loss due to the disease or falls, and (d) transportation. For estimating productivity loss using the human capital method, each individual will be assessed using a 'market value' based on the future earning of the individual if he/she was in good health status.

Data collection process One research assistant will be recruited to conduct the assessments and will be supervised by the primary investigator. All the assessments and surveys will be carried out at the Hong Kong Polytechnic University campus. For participants expressing difficulty in reaching the venue, the assessments will be carried out at their residence. After explaining the purposes, procedures and potential risks of the study, participants will complete the informed consent prior to data collection. The cost data sheet is a 52 items self-reported spreadsheet to be completed by the patients or their caregivers (Appendix 1). The disease severity of the participants will be assessed by the research assistant, trained and supervised by the PI. Other than the assessor, stand-by assistance will be provided to ensure safety. The total time required for the three tests was less than an hour.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling participants with a confirmed diagnosis of Parkinson's disease
* both genders
* any age
* who are residing in Hong Kong.

Exclusion Criteria:

* are wheelchair-bound or bed-ridden,
* have atypical Parkinson's syndrome and
* other associated major illness such as stroke.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community-dwelling participants with a confirmed diagnosis of Parkinson's disease of both genders of any age and who are residing in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Healthcare cost | Ongoing assessment from day 1 until 12 months
  We will estimate both direct and indirect cost using the self-reported questionnaires available in both English and Chinese languages. The following criteria were used to choose the individual items under direct and indirect costs: relevance to Parkinson's disease, relevance to falls and consequences of falls, how quantifiable the items are, based on the commonly estimated items in similar economic, and to the extent to which the item reflects and impacts the quality of life of people with Parkinson's disease.

SECONDARY OUTCOMES:
Number of falls | Day 1 (T1), 6 months (T2) and 12 months (T3)
  In this study, we define falls as a rapid uncontrolled change from sitting or upright position to the reclining of coming to the ground, and 'frequent fallers' as those who fell 5 or more times per twelve months, 'infrequent fallers' as those having less than 4 falls and 'non-fallers with those having no falls
MDS-UPDRS | Day 1 (T1), 6 months (T2) and 12 months (T3)
  MDS-UPDRS: is a measure of severity due to Parkinson's disease. The scale is scored between 0 and 199, where 0 indicates no disability and 199 implies to maximal disability due to the disease. The severity is scored across 5 segments including (i) mental, behaviour and mood, (ii) activities of daily living, (iii) motor examination, (iv) modified Hoehn and Yahr Scale and (v) Schwab and England ADL scale. In this study, we will use the simplified Chinese version of the scale
Hoehn and Yahr scale | Day 1 (T1), 6 months (T2) and 12 months (T3)
  Hoehn and Yahr scale: is a measure of the level of disability and symptom progress due to Parkinson's disease. The scale classifies the patient from stage 0 (no signs) to stage 5 (bedridden or wheelchair-bound).
MiniBESTest | Day 1 (T1), 6 months (T2) and 12 months (T3)
  MiniBESTest: is a generic measure of balance and falls risk prediction in neurological disorders. The BESTest is found to be valid and reliable in people with PD. The scale measures anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait. The scale has 14 items and is scored out of 28 with a lower score indicating poor balance and postural control
Falls Efficacy Scale International (FES-I) | Day 1 (T1), 6 months (T2) and 12 months (T3)
  Falls Efficacy Scale International (FES-I): is a self-reported measure for assessing the fear of falls among community-dwelling older adults. The scale has 16 items scored between 1 and 4. The scale has a minimum score of 16 indicating no concerns of falls and a maximum score of 46 indicating maximal falls concern. The FES-I is found to be a valid measure for estimating the falls risk prediction among people with Parkinson's disease
Activities-specific Balance Confidence (ABC) scale | Day 1 (T1), 6 months (T2) and 12 months (T3)
  Activities-specific Balance Confidence (ABC) scale: is a generic, self-reported measure for estimating the balance confidence. The scale has 16 items, each rated between 0% indicating no confidence and 100% indicating complete confidence in the activity. The higher the score obtained better the balance performance. The ABC os found to be valid and reliable for assessing balance among people with Parkinson's disease
Short-form Health survey (SF-36) | Day 1 (T1), 6 months (T2) and 12 months (T3)
  Short-form Health survey (SF-36): The Short Form (36) Health Survey (SF-36) will be used to measure the quality of life. The scale is scored between 0 and 100 across the eight domains, with 0 indicating the worst health and 100 indicating the best health status possible. The Chinese version of SF-36 was used in the current work. This version exhibits satisfactory convergent and discriminant validities

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J Winser, PhD, Principal Investigator — The Hong Kong Polytechnic Universit
Locations (2):
- Hong Kong (2):
  - The Hong Kong Polytechnic University, Hung Hom, Kowloon
  - Prince of Wales Hospital, Shatin

IPD SHARING:
Plan to Share IPD: No
The personnel identification of the included participants will not be revealed. The study-related data will be expressed using a unique identification ID number. Personnel identifications such as names or photos will not be identified in public events such as conference presentations.